CLINICAL TRIAL: NCT01575652
Title: Effects of Angiotensin Converting Enzyme Inhibitors on Peritoneal Protein Loss and Solute Transport in Peritoneal Dialysis Patients
Brief Title: Effects of Aceis on Peritoneal Protein Loss and Solute Transport in pd Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turkish Nephrology Association (Other)
Responsible Party: Principal Investigator, taner basturk, Principle Investigator, Turkish Nephrology Association
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D-11-00212R1
Record Dates: First submitted 2012-04-04; First posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Disorders Associated With Peritoneal Dialysis
Keywords: peritoneal dialysis; protein losses
MeSH Terms: interventions — Perindopril; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE-I (Active Comparator): Group using ACEIs
  Interventions: Other: Group using angiotensin converting enzyme inhibitor
- ACE-I, 2 (No Intervention): group not using ace-i
  Interventions: Other: Group not using angiotensin converting enzyme inhibitor

INTERVENTIONS:
Other: Group using angiotensin converting enzyme inhibitor — Measurement of peritoneal protein loss level with use of ACEIs
  Other Names: Perindopril; Lisinopril
  Arms: ACE-I
Other: Group not using angiotensin converting enzyme inhibitor — Measurement of peritoneal protein loss level without usage of ACEIs
  Arms: ACE-I, 2

SUMMARY:
The objective of this study was to examine the effects of angiotensin converting enzyme inhibitors on peritoneal membrane transport, peritoneal protein loss, and proteinuria in peritoneal dialysis patients.

DETAILED DESCRIPTION:
This prospective cohort study was conducted at the Unit of Nephrology of Sisli Etfal Education and Research Hospital, Istanbul, Turkey. Prior to subject recruitment, the study protocol was reviewed and approved by the local ethics committee, in accordance with the ethical principles for human investigations, and written informed consents were obtained from all patients. Between june 2008 and january 2009, 54 age and gender matched continuous ambulatory peritoneal dialysis (CAPD) patients were included in the study consecutively.

Patients were divided into 2 groups according to decision of the physician; group 1 (n=34) was consisted of patients treated with ACE-Is and group 2 (n=30) was not treated with ACEs. The inclusion criteria were chronic PD patients between 18 and 85 years who had not received any antihypertensive drugs within prior 12 months. All patients were on standard CAPD program (2-2.5 L; 4 exchanges/day). Icodextrin is not used. The exclusion criteria were as follows; patients who had a history of antihypertensive treatment with ACE-Is or angiotensin-receptor blockers or aldosterone antagonists for prior 12 months from the study time; intolerance to the ACE-Is; CAPD-related peritonitis within 6 months prior to or during the study period; history of malignant hypertension or hypertensive encephalopathy or cerebrovascular accident within the 6 months prior to the study; chronic liver diseases, and recent acute illness and/or history of any overt chronic inflammatory disease.

Demographic variables including etiology of CKD, age, and gender were obtained from patients' clinic charts. All blood samples were taken after 10 hours of overnight fasting. Serum urea, creatinine, and albumin levels were analyzed. Creatinine clearance [(CCr) dialysate, urine, and total], Kt/V (dialysate, urine, and total) were calculated weekly. Daily volumes (UF), 24-hour protein, and albumin losses (dialysate, urine) were recorded also. Parameters at the beginning of study and at the end of 6th month were evaluated. During the study, the dialysis regime remained same in all patients. In both groups, investigators analyzed blood, 24-hour urine (in patients with residual diuresis >100mL daily), peritoneal effluent fluid at 4 hours' and 24 hours' dwell time. Peritoneal effluent fluid at 24 hours' dwell time was used to determine total protein, albumin, and at 24 hours' dwell time to determine urea and creatinine. The urea kinetic test in closest time proximity to the PET was used in the analysis.

After the subject had rested in the supine position for at least 15 minutes blood pressure was measured with a standard mercury sphyngomanometer for the three times with the half of a cuff around the right arm. Patients' blood pressure measurements were performed on a regular basis every month. The mean values were calculated. All patients received standard 35-cal/kg/day carbohydrate, 1-2 g/kg/day protein, and salt restricted diet. Patients did not use essential amino acid and peritoneal dialysis solutions containing amino acids. Serum urea, creatinine, and albumin levels were assessed by enzymatic colorimetric assay. Dialysate adequacy (Kt/V urea: dialysis and residual), and peritoneal transport (4-hour D/PCr) were measured using standard procedures (PD Adequest 1.4, 1994: Baxter Healthcare Corporation, Deerfield, IL, U.S.A.). Dialysate albumin loss was measured with the Bromo Cresol Green (BCG) method. Dialysate total protein loss was measured by the Biuret method. Urine protein concentration was determined by an immunoturbidimetric method.

Statistical analysis was carried out using the SPSS 13.0 software package (SPSS Inc, Chicago, IL, USA). Kolmogorov-Smirnov tests were used to test the normality of data distribution. Data were expressed as arithmetic means and standard deviations. Chi-square test was used to compare the categorical variables between groups. Independent sample T-test and Mann-Whitney U tests were used respectively between groups in normally and abnormally distributed continuous variables. Paired t-test and Wilcoxon signed-rank tests were used to analyze changes within each group. Two-sided p value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* chronic peritoneal dialysis First paragraph.
* 18- 55 years
* no antihypertensive drug usage prior 12 months

Exclusion Criteria:

* usage of antihypertensives prior 12 months
* intolerance to the ace-i
* CAPD related peritonitis prior 6 months or during the study time
* history of malignant hypertension or hypertensive encephalopathy or cerebrovascular accident within the 6 months prior to the study
* chronic liver diseases
* recent acute illness and/or history of any overt chronic inflammatory disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
degree of peritoneal protein loss | 6 months
  measurement of peritoneal protein loss after 6 months treatment of acei

CONTACTS AND LOCATIONS:
Overall Officials: taner basturk, MD, Principal Investigator — Sisli Etfal training and Education Hospital

REFERENCES:
- [Result] Rubin J, Adair C, Barnes T, Bower J. Dialysate flow rate and peritoneal clearance. Am J Kidney Dis. 1984 Nov;4(3):260-7. doi: 10.1016/s0272-6386(84)80103-1. PMID 6496469
- [Result] Krediet RT, Zuyderhoudt FM, Boeschoten EW, Arisz L. Peritoneal permeability to proteins in diabetic and non-diabetic continuous ambulatory peritoneal dialysis patients. Nephron. 1986;42(2):133-40. doi: 10.1159/000183652. PMID 3945351
- [Result] Davies SJ, Bryan J, Phillips L, Russell GI. Longitudinal changes in peritoneal kinetics: the effects of peritoneal dialysis and peritonitis. Nephrol Dial Transplant. 1996 Mar;11(3):498-506. PMID 8671821
- See also: fda approval of perindopril — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Overview&DrugName=PERINDOPRIL%20ERBUMINE
- See also: fda approval of lisinopril — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.Overview&DrugName=LISINOPRIL